CLINICAL TRIAL: NCT05691972
Title: A Randomized, No-treatment-controlled, Evaluator-blinded, Multi-center Study to Evaluate the Effectiveness and Safety of Restylane Contour in the Treatment of Temple Hollowing
Brief Title: Effectiveness and Safety of Restylane Contour in the Treatment of Temple Hollowing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43USTH2201
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Temporal Hollowing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment (Experimental)
  Interventions: Device: Restylane Contour
- Control (No Intervention)

INTERVENTIONS:
Device: Restylane Contour — a sterile, biodegradable, transparent gel of nonanimal cross-linked HA (20 mg/mL) with the addition of lidocaine hydrochloride (3 mg/mL)
  Arms: Treatment

SUMMARY:
This is a randomized, no-treatment-controlled, evaluator-blinded, multi-center study to evaluate the effectiveness and safety of Restylane® Contour in correction of temple hollowing.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant, non-breastfeeding females, 22 years of age or older
* Intent to undergo treatment for correction of temple hollowing

Exclusion Criteria:

* Known/previous allergy or hypersensitivity to any injectable hyaluronic acid (HA) gel or to gram positive bacterial proteins
* Known/previous allergy or hypersensitivity to local anesthetics, e.g., lidocaine or other amide-type anesthetics or nerve blocking agents (if intended to be used for that subject)
* Previous facial surgery (e.g., facelift) above the level of the horizontal line from subnasale that in the Treating Investigator´s opinion could interfere with the study safety and/or effectiveness assessments
* Any previous aesthetic procedures or implants
* Recurrent temporal headaches such as temporal tendinitis migraine. Have a history of migraines or frequent headaches, as determined by the (Treating) Investigator, that could interfere with the study safety and/or effectiveness assessments

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
Responder rate based on the Blinded Evaluators' live assessment of the GTVDS | Baseline to 3 months

SECONDARY OUTCOMES:
Responder rates, as assessed by the Blinded Evaluator at 6, 9 and 12 months after baseline for the treatment group | 6,9,12 months after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Galderma R&D
Locations (15):
- United States (15):
  - Galderma Research Site, Phoenix, Arizona
  - Galderma Research Site, Encino, California
  - Galderma Research Site, Los Angeles, California
  - Galderma Research Site, Redondo Beach, California
  - Galderma Research Site, Solana Beach, California
  - Galderma Research Site, Vista, California
  - Galderma Research Site, Washington D.C., District of Columbia
  - Galderma Research Site, Adventura, Florida
  - Galderma Research Site, Boynton Beach, Florida
  - Galderma Research Site, Coral Gables, Florida
  - Galderma Research Site, New Orleans, Louisiana
  - Galderma Research Site, New York, New York
  - Galderma Research Site, Chapel Hill, North Carolina
  - Galderma Research Site, Wilmington, North Carolina
  - Galderma Research Site, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No